CLINICAL TRIAL: NCT07138508
Title: Oral Nicorandil for Prevention of No Reflow Phenomenon in Anterior STEMI Patients Undergoing PPCI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Misr University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MS188/2024
Record Dates: First submitted 2025-07-05; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: No Reflow Phenomenon; Anterior STEMI
Keywords: Nicorandil; No reflow; Anterior STEMI
MeSH Terms: conditions — No-Reflow Phenomenon | interventions — Nicorandil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome of the study was assessed by an interventional cardiologist blind to group allocation:
  Final TIMI Final MBG
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Has not received oral nicorandil
- Treatment (Active Comparator): Received 20mg of oral nicorandil
  Interventions: Drug: Nicorandil 20mg

INTERVENTIONS:
Drug: Nicorandil 20mg — Oral nicorandil 20mg
  Arms: Treatment

SUMMARY:
Aim of the study is to Investigate the potential role of oral nicorandil in preventing the No reflow phenomenon in anterior ST-segment elevation myocardial infarction (STEMI) patients undergoing percutaneous coronary intervention (PPCI).

Assess whether nicorandil, a potassium channel activator, can effectively enhance myocardial perfusion in this specific clinical context.

* In a randomized controlled trial study
* All recruited patients were randomized to either the treatment or control group in a ratio of 1:1 using a computer-generated randomization sequence in relation to the order of participation in the study. Patients fulfilling the inclusion criteria and consenting to participate in the study were recruited.

DETAILED DESCRIPTION:
This is a randomized, controlled clinical trial designed to evaluate the efficacy of a single oral dose of nicorandil in preventing the no-reflow phenomenon in patients with anterior ST-segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PPCI).

Study Setting:

The study is conducted at the Cardiology Departments of Ain Shams University Hospitals and Misr University for Science and Technology Hospitals.

Study intervention:

Group A (Study Group): Receives a single oral dose of nicorandil 20 mg prior to PPCI.

Group B (Control Group):Undergoes PPCI without receiving nicorandil.

Randomization and Sampling:

Patients meeting the inclusion criteria and providing informed consent are randomized using a computer-generated sequence to ensure unbiased allocation. A total of 300 patients enrolled, with 150 patients per group.

Ethical Considerations:

Ethical approval has been obtained from the Ethical Committee Board of Ain Shams University, and the study is conducted in accordance with the principles of the Declaration of Helsinki. Written informed consent is obtained from all participants either in the emergency department or catheterization laboratory prior to the intervention.

Study Procedures:

All enrolled patients undergo:

Comprehensive Clinical Evaluation:

Detailed history with emphasis on coronary artery disease (CAD) risk factors:

* Age
* Sex
* Diabetes Mellitus (DM)
* Hypertension (HTN)
* Family history of ischemic heart disease (IHD)
* Dyslipidemia
* Chronic kidney disease (CKD)
* Smoking status
* Clinical presentation and functional status using the Killip classification.
* Vital signs monitoring.

Electrocardiogram (ECG):

Standard 12-lead ECG obtained on first medical contact to confirm STEMI diagnosis.

All PCI procedures are performed by experienced interventional cardiologists using standardized protocols for anterior STEMI intervention.

Data Collection and Assessments:

Angiographic Data:

TIMI flow grade is assessed post-PCI by two independent interventional cardiologists blinded to treatment allocation to objectively evaluate coronary flow.

Echocardiographic Assessment:

Transthoracic echocardiography (TTE) is performed after PCI and prior to hospital discharge.

Left ventricular ejection fraction (LVEF) is measured using the modified Simpson's method by an independent echocardiographer blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients diagnosed with anterior ST-segment elevation myocardial infarction (STEMI).
* Individuals scheduled for percutaneous coronary intervention (PPCI).
* Presence of risk factors or indications for preventing the No reflow phenomenon.
* Willingness and ability to comply with the study protocol.
* Ability to provide informed consent for participation in the study.

Exclusion Criteria:

* Known allergic reaction to oral nicorandil.
* Concomitant use of medications that may interact with nicorandil.
* Presence of contraindications to oral nicorandil such as hypotension, hepatic or renal impairment
* Need for emergent coronary artery bypass grafting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
No reflow using angiographic criteria | Intra procedural
  Incidence of No reflow

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 1 week from procedure
  Incident of stroke, reinfarction, arrhythmia and cardiac arrest were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
IPD data will shared after obtaining publication acceptance

DOCUMENTS (1):
  • Informed Consent Form (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT07138508/ICF_000.pdf